CLINICAL TRIAL: NCT03062891
Title: Sleep Treatment Outcome Predictors: A Pilot Study (STOP-pilot)
Acronym: STOP-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Goldsmiths, University of London (Other); Queen Mary University of London (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP-0001-PILOT
Record Dates: First submitted 2016-12-05; First posted 2017-02-24 (Actual); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2017-01

CONDITIONS: Sleep Problem
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online CBT for insomnia (Experimental): CBT participants will receive six weekly sessions delivered by an animated 'virtual therapist' (The Prof) via the online platform 'Sleepio'. The programme comprises a fully automated media-rich web application, driven dynamically by baseline, adherence, performance and progress data, and provides additional access to elements such as an online library with background information, a community of fellow users, and support, prompts and reminders sent by e-mail.
  CBT content was consistent with the literature (4) and covered behavioral (e.g., sleep restriction, stimulus control) and cognitive (e.g., putting the day to rest, thought restructuring, imagery, articulatory suppression, paradoxical intention, mindfulness) strategies, as well as additional relaxation strategies (progressive muscle relaxation and autogenic training) and advice on lifestyle and bedroom factors (sleep hygiene). The intervention was based upon a previously validated manual (4).
  Interventions: Procedure: Online CBT for insomnia
- Puzzles (No Intervention): Each week participants will be sent a puzzle to complete online (e.g. logic puzzles, crosswords etc). The puzzles have been designed to be cognitively engaging and take a similar amount of time to one session of Sleepio (20-25 minutes).

INTERVENTIONS:
Procedure: Online CBT for insomnia — See CBT arm description for information about the CBT intervention. More details can be found in source 4 in the reference list.
  Arms: Online CBT for insomnia

SUMMARY:
Insomnia occurs frequently causing a substantial burden to society (1). Historically, insomnia has been considered as secondary to a handful of other psychiatric disorders, such as depression and anxiety - but it is now clear that this disorder is associated with a wide range of psychiatric conditions and may actually precede and predict their development and severity (e.g. 2). Treating insomnia has been posited to hold the promise of reducing or preventing the development of co-morbid problems - although this possibility needs to be rigorously tested.

Cognitive behavioural therapy (CBT) is an effective treatment for disturbed sleep, specifically insomnia, in adults (3) and is recommended by NICE for the management of long-term sleep problems. This treatment is more accessible than ever before given recent ground-breaking internet initiatives - such as the Sleepio programme (see: https://www.sleepio.com/home/), which was developed by one of the collaborators (Colin Espie) and has yielded encouraging results (4).

Despite the importance of CBT for treating disturbed sleep and the finding that it leads to a good outcome for the majority of sufferers, some people fail to respond to this treatment. For example, research cited on the Sleepio website notes that around 70% of those with even very long term sleep difficulties experience long-term improvements from the treatment, meaning that 30% do not (see 4). Understanding more about who does and does not respond holds the promise of improving or tailoring treatments for insomnia.

The study proposed here builds on recent work by one of the researchers who has been exploring demographic (5), clinical (e.g. 6) and most uniquely genetic (e.g. 7); and epigenetic (e.g. 8) predictors of psychological treatment response (coining the term Therapygenetics, see, 7). While these predictors are individually only likely to explain a small proportion of the variance of treatment outcome, understanding these multiple risks and their interaction is the best way to consider this issue. The study addressed here is a pilot study, necessary to demonstrate feasibility of utilising a sleep intervention application in an unselected sample of young adults, prior to applying for grant funding to undertake a larger but similar behavioural genetics study in the future.

The main aim of this pilot study is to test the feasibility of the study design, by investigating whether unselected participants show an improvement in sleep quality after taking the intervention. Participation and drop out rates as well acceptability of the intervention in a non-clinical population will also be investigated.

Research Questions:

1. Does the online CBT intervention improve sleep quality in a non-clinical, unselected sample?
2. How feasible is it to run this study on a non-clinical sample? This will include investigating response rate, participant drop-out, and treatment accessibility.

   The investigators will also offer perform preliminary investigations into:
3. Does improving sleep quality have implications for associated phenotypes? Specifically the investigators will examine symptoms of anxiety, depression, attention-deficit hyperactivity disorder (ADHD), psychosis, and well-being.
4. Which demographic, clinical, genetic, and epigenetic factors predict treatment outcome for sleep problems?

Research questions 3) and 4) will be primary aims in the main study, but will constitute secondary aims in the pilot study as there won't be the statistical power to fully address these questions.

ELIGIBILITY:
Inclusion

* Female
* Aged 18 plus
* Psychology student (undergraduate or postgraduate) at one of three London universities involved in the study.

Exclusion

* Male
* Under 18
* Not a psychology student (undergraduate or postgraduate) at one of three London universities involved in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Gregory, PhD, Principal Investigator — Goldsmiths, University of London
Locations (3):
- United Kingdom (3):
  - Queen Mary, University of London, London
  - Goldsmiths, University of London, London
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund PA, Coulouvrat C, Hajak G, Roth T, Shahly V, Shillington AC, Stephenson JJ, Walsh JK. Insomnia and the performance of US workers: results from the America insomnia survey. Sleep. 2011 Sep 1;34(9):1161-71. doi: 10.5665/SLEEP.1230. PMID 21886353
- [Background] Harvey AG. Insomnia: symptom or diagnosis? Clin Psychol Rev. 2001 Oct;21(7):1037-59. doi: 10.1016/s0272-7358(00)00083-0. PMID 11584515
- [Background] Morin CM, Bootzin RR, Buysse DJ, Edinger JD, Espie CA, Lichstein KL. Psychological and behavioral treatment of insomnia:update of the recent evidence (1998-2004). Sleep. 2006 Nov;29(11):1398-414. doi: 10.1093/sleep/29.11.1398. PMID 17162986
- [Background] Espie CA, Kyle SD, Williams C, Ong JC, Douglas NJ, Hames P, Brown JS. A randomized, placebo-controlled trial of online cognitive behavioral therapy for chronic insomnia disorder delivered via an automated media-rich web application. Sleep. 2012 Jun 1;35(6):769-81. doi: 10.5665/sleep.1872. PMID 22654196
- [Background] Hudson JL, Lester KJ, Lewis CM, Tropeano M, Creswell C, Collier DA, Cooper P, Lyneham HJ, Morris T, Rapee RM, Roberts S, Donald JA, Eley TC. Predicting outcomes following cognitive behaviour therapy in child anxiety disorders: the influence of genetic, demographic and clinical information. J Child Psychol Psychiatry. 2013 Oct;54(10):1086-94. doi: 10.1111/jcpp.12092. Epub 2013 Jun 18. PMID 23772677
- [Background] Hudson JL, Keers R, Roberts S, Coleman JR, Breen G, Arendt K, Bogels S, Cooper P, Creswell C, Hartman C, Heiervang ER, Hotzel K, In-Albon T, Lavallee K, Lyneham HJ, Marin CE, McKinnon A, Meiser-Stedman R, Morris T, Nauta M, Rapee RM, Schneider S, Schneider SC, Silverman WK, Thastum M, Thirlwall K, Waite P, Wergeland GJ, Lester KJ, Eley TC. Clinical Predictors of Response to Cognitive-Behavioral Therapy in Pediatric Anxiety Disorders: The Genes for Treatment (GxT) Study. J Am Acad Child Adolesc Psychiatry. 2015 Jun;54(6):454-63. doi: 10.1016/j.jaac.2015.03.018. Epub 2015 Apr 1. PMID 26004660
- [Background] Eley TC, Hudson JL, Creswell C, Tropeano M, Lester KJ, Cooper P, Farmer A, Lewis CM, Lyneham HJ, Rapee RM, Uher R, Zavos HM, Collier DA. Therapygenetics: the 5HTTLPR and response to psychological therapy. Mol Psychiatry. 2012 Mar;17(3):236-7. doi: 10.1038/mp.2011.132. Epub 2011 Oct 25. No abstract available. PMID 22024766
- [Background] Roberts S, Lester KJ, Hudson JL, Rapee RM, Creswell C, Cooper PJ, Thirlwall KJ, Coleman JR, Breen G, Wong CC, Eley TC. Serotonin transporter [corrected] methylation and response to cognitive behaviour therapy in children with anxiety disorders. Transl Psychiatry. 2014 Sep 16;4(9):e444. doi: 10.1038/tp.2014.83. PMID 25226553
- [Background] Vgontzas AN, Fernandez-Mendoza J, Liao D, Bixler EO. Insomnia with objective short sleep duration: the most biologically severe phenotype of the disorder. Sleep Med Rev. 2013 Aug;17(4):241-54. doi: 10.1016/j.smrv.2012.09.005. Epub 2013 Feb 16. PMID 23419741
- [Derived] Denis D, Poerio GL, Derveeuw S, Badini I, Gregory AM. Associations between exploding head syndrome and measures of sleep quality and experiences, dissociation, and well-being. Sleep. 2019 Feb 1;42(2). doi: 10.1093/sleep/zsy216. PMID 30544141
- [Derived] Denis D, Eley TC, Rijsdijk F, Zavos HMS, Keers R, Espie CA, Luik AI, Badini I, Derveeuw S, Romero A, Hodsoll J, Gregory AM. Sleep Treatment Outcome Predictors (STOP) Pilot Study: a protocol for a randomised controlled trial examining predictors of change of insomnia symptoms and associated traits following cognitive-behavioural therapy for insomnia in an unselected sample. BMJ Open. 2017 Dec 1;7(11):e017177. doi: 10.1136/bmjopen-2017-017177. PMID 29196479
- See also: Sleepio website - the online CBT platform used in the study — http://www.sleepio.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 240 participants gave informed consent. After consent, participants were required to complete the baseline assessments before being assigned to a group. A total of 41 participants did not fill out this survey despite consenting, meaning a total of 199 participants were assigned to a group.
Period: Overall Study
Arm/Group | Online CBT for Insomnia | Puzzles
Started | 99 | 100
Mid-intervention | 68 | 74
End of Intervention | 67 | 78
Followup | 47 | 62
Completed | 47 | 62
Not Completed | 52 | 38
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 50 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online CBT for Insomnia | Puzzles | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.73 (2.94) | 20.22 (5.69) | 20.22 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 100 | 199
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arab | 4 | 1 | 5
  Asian or Asian British | 10 | 20 | 30
  Black or Black Britsh | 6 | 5 | 11
  Mixed ethnicity | 6 | 8 | 14
  Other | 5 | 5 | 10
  White | 43 | 41 | 84
  Selected more than one ethnicity | 25 | 19 | 44
  Prefer not to say | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 99 | 100 | 199
Insomnia symptoms [Mean (Standard Deviation); unit: units on a scale] — The scale used was the Sleep Condition Indicator (SCI). This scale has a theoretical range of 0-32. A higher score indicates fewer insomnia symptoms.
  units on a scale | 19.70 (6.56) | 20.22 (6.53) | 19.97 (6.53)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Insomnia Symptoms Following Online CBT
Description: Changes in insomnia symptoms as assessed by scores on the Sleep Condition Indicator (SCI). This pilot aims to establish the distributional properties of individual differences in change score on this measure. The scale has a theoretical range of 0-32. A higher score indicates fewer insomnia symptoms. Therefore a positive change score (>0) indicates fewer insomnia symptoms at the end of the intervention compared to baseline. A negative score (<0) indicates more symptoms at the end of the itnervention compared to baseline.
Time Frame: Change from baseline to 3 weeks, 6 weeks, and 6 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 67 | 74
score on a scale
  3 weeks | 2.98 [1.93 to 4.04] | 1.26 [-0.06 to 2.57]
  6 weeks | 4.69 [3.82 to 5.99] | 2.34 [1.00 to 3.67]
  6 months | 4.89 [3.08 to 6.69] | 2.05 [0.31 to 3.79]

2. Primary Outcome: Improvement in Sleep Quality Following Online CBT
Description: Changes in sleep quality as assessed by scores on the Pittsburgh Sleep Quality Index (PSQI). This pilot aims to establish the distributional properties of individual differences in change score on this measure. The scale has a theoretical range of 0-21. The change score reflects the change in symptoms at each assessment compared with baseline. Higher scores on the indicate worse sleep quality. Therefore for the change score, a positive value indicates worse sleep quality at the assessment time period compared to baseline. A negative value indicates better sleep quality at the assessment time period compared to baseline.
Time Frame: Change from baseline to 3 weeks, 6 weeks, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 67 | 74
score on a scale
  3 weeks | -0.71 (3.32) | -0.47 (3.47)
  6 weeks | -1.92 (3.35) | -1.11 (2.94)
  6 months | 0 (4.41) | -1.56 (3.53)

3. Primary Outcome: Treatment Acceptability Mid-intervention
Description: Acceptability of the CBT-I in an unselected sample will be assessed, and measured using an adapted version of the Treatment Acceptability Questionnaire (TAQ) suitable for use with an online therapist. The TAQ has a theoretical range of 6-42, with a higher score indicating higher levels of treatment acceptability.
Time Frame: 3 weeks
Population: Treatment acceptability was only measured in the Online CBT for insomnia group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 68 | 0
score on a scale | 29.96 (3.79) |

4. Primary Outcome: Treatment Acceptability at the End of the Intervention
Description: as for outcome 3
Time Frame: 6 weeks
Population: Treatment acceptability was only measured in the Online CBT for insomnia group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 67 | 0
score on a scale | 33.61 (4.82) |

5. Primary Outcome: Change in Treatment Acceptability During the Intervention
Description: Change in treatment acceptability across the CBT-I treatment will be assessed, through changes in the score on the Treatment Acceptability Scale. Acceptability of the CBT-I in an unselected sample will be assessed, and measured using an adapted version of the Treatment Acceptability Questionnaire (TAQ) suitable for use with an online therapist. The TAQ has a theoretical range of 6-42, with a higher score indicating higher levels of treatment acceptability. Therefore a positive change score means an improvement in treatment acceptability, whereas a negative change score indicates a reduction in treatment acceptability.
Time Frame: Change from baseline to 3 weeks and 6 weeks
Population: Treatment acceptability was only assessed in the Online CBT for insomnia group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 67 | 0
score on a scale | 3.65 (3.98) |

6. Primary Outcome: Attrition Rate
Description: Drop-out rate will be assessed as the percentage of those who consented to take part in the study who did not complete the study.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
percentage of participants | 47 | 62

7. Secondary Outcome: Predictors of Treatment Outcome - Anxiety
Description: Anxiety as a predictor of response to treatment outcome, as measured using the Trait State Anxiety Index. The theoretical range is 20-80, and a higher score indicates more anxiety symptoms at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 49.93 (10.64) | 47.53 (9.92)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline anxiety symptoms and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .572, Regression, Linear; Slope = 0.54, 95% CI 2-sided [-1.33 to 2.40]

8. Secondary Outcome: Predictors of Treatment Outcome - Depression
Description: Anxiety as a predictor of response to treatment outcome, as measured using the Mood and Feelings Questionnaire. The theoretical range is 0-26, and a higher score indicates more anxiety symptoms at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 10.09 (6.71) | 8.65 (6.27)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline depression symptoms and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .934, Regression, Linear; Slope = 0.08, 95% CI 2-sided [-1.82 to 1.98]

9. Secondary Outcome: Predictors of Treatment Outcome - Attentional Problems
Description: Attentional problems as a predictor of response to treatment outcome, as measured using the ADHD symptoms questionnaire. The theoretical range is 1-54, and a higher score indicates more attentional problems at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 21.47 (11.69) | 22.09 (11.62)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between attentional problems and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .253, Regression, Linear; Slope = 1.07, 95% CI 2-sided [-0.76 to 2.89]

10. Secondary Outcome: Predictors of Treatment Outcome - Psychotic Experiences
Description: Psychotic experiences as a predictor of response to treatment outcome, as measured using the Specific Psychotic Experiences Questionnaire. Subsacles measuring paranoia (theoretical range 0-25), hallucinations (theoretical range 0-25), and cognitive disorganization (0-5) were used. On all subscales, a higher score indicates more psychotic experiences at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Paranoia | 6.66 (5.76) | 6.43 (5.20)
  Hallucinations | 3.03 (3.71) | 2.02 (2.55)
  Cognitive disorganization | 3.19 (1.55) | 3.33 (1.55)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline paranois and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .215, Regression, Linear; Slope = 1.20, 95% CI 2-sided [-0.70 to 3.10]
Statistical Analysis 2: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline hallucinations and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .254, Regression, Linear; Slope = 1.14, 95% CI 2-sided [-0.83 to 3.11]
Statistical Analysis 3: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline cognitive disorganization and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .778, Regression, Linear; Slope = -0.27, 95% CI 2-sided [-2.13 to 1.59]

11. Secondary Outcome: Predictors of Treatment Outcome - Positive Mental Health
Description: Positive mental health as a predictor of response to treatment outcome, as measured using the Positive Mental Health Scale. The theoretical range is 1-36, and a higher score indicates higher levels of positive mental health at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 26.00 (6.44) | 26.64 (5.76)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline positive mental health and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .800, Regression, Linear; Slope = -0.25, 95% CI 2-sided [-2.16 to 1.67]

12. Secondary Outcome: Predictors of Treatment Outcome - Stress
Description: Stress as a predictor of response to treatment outcome, as measured using the Perceived Stress Scale. The theoretical range is 5-50, and a higher score indicates more perceived stress at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 20.14 (6.82) | 20.05 (6.12)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline perceived stress and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .525, Regression, Linear; Slope = 0.59, 95% CI 2-sided [-1.25 to 2.44]

13. Secondary Outcome: Predictors of Treatment Outcome - Threatening Life Events
Description: Threatening life events as a predictor of response to treatment outcome, as measured using the List of Threatening Events. The theoretical range is 0-24, and a higher score indicates more exposure to threatening events in the 12 months preceeding baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 2.57 (2.31) | 2.72 (2.69)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the interaction between baseline threatening life events and group on the change in insomnia symptoms across the intervention. The results of the interaction are reported here; Test type: Superiority; p = .140, Regression, Linear; Slope = 1.30, 95% CI 2-sided [-0.43 to 3.03]

14. Secondary Outcome: Changes in Scores on Associated Phenotypes - Anxiety
Description: Anxiety symptoms, measured using the State Trait Anxiety Index. The theoretical range is 20-80, and a higher score indicates more anxiety symptoms at baseline.
Time Frame: 3 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Mid intervention | 46.68 (11.86) | 46.58 (10.26)
  End of intervention | 44.57 (11.20) | 45.32 (10.07)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in anxiety symptoms across the intervention period; Test type: Superiority; p = .030, Generalized estimating equation; Slope = -2.58, 95% CI 2-sided [-4.90 to -0.25]

15. Secondary Outcome: Changes in Scores on Associated Phenotypes - Depression
Description: Depression symptoms, as measured using the Trait State Anxiety Index. The theoretical range is 0-26, and a higher score indicates more depression symptoms.
Time Frame: 3 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Mid intervention | 8.70 (7.20) | 8.00 (7.01)
  End of intervention | 6.91 (5.73) | 6.51 (5.87)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in depression symptoms across the intervention period; Test type: Superiority; p = .456, Generalized estimating equation; Slope = -0.63, 95% CI 2-sided [-2.24 to 1.01]

16. Secondary Outcome: Changes in Scores on Associated Phenotypes - Attentional Problems
Description: Attentional problems, as measured using the ADHD symptoms questionnaire. The theoretical range is 1-54, and a higher score indicates more attentional problems.
Time Frame: 3 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale | 16.51 (10.53) | 18.53 (13.33)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes attentional problems across the intervention period; Test type: Superiority; p = .110, Generalized estimating equation; Slope = -2.34, 95% CI 2-sided [-5.21 to 0.53]

17. Secondary Outcome: Changes in Scores on Associated Phenotypes - Psychotic Experiences
Description: Psychotic experiences, as measured using the Specific Psychotic Experiences Questionnaire. Three subscales measuring paranoia (theoretical ragne 0-25), hallucinations (0-25), and cognitive disorganization (0-5) were used. On all subscales, a higher score equals more frequent experiences
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Paranoia | 4.59 (5.77) | 6.07 (5.92)
  Hallucinations | 1.59 (3.24) | 1.31 (2.42)
  Cognitive disorganization | 2.65 (1.89) | 3.07 (1.52)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in psychotic experiences (paranoia) across the intervention period; Test type: Superiority; p = .041, Generalized estimating equations; Slope = -1.69, 95% CI 2-sided [-3.31 to -0.07]
Statistical Analysis 2: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in psychotic experiences (hallucinations) across the intervention period; Test type: Superiority; p = .531, Generalized estimating equation; Slope = -0.22, 95% CI 2-sided [-0.92 to 0.48]
Statistical Analysis 3: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in psychotic experiences (cognitive disorganization) across the intervention period; Test type: Superiority; p = .130, Generalized estimating equation; Slope = -0.37, 95% CI 2-sided [-0.84 to 0.11]

18. Secondary Outcome: Changes in Scores on Associated Phenotypes - Positive Mental Health
Description: Positive mental health, as measured using the Positive Mental Health Scale. The theoretical range is 1-36, and a higher score indicates higher levels of positive mental health.
Time Frame: 3 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Mid intervention | 25.39 (7.01) | 26.46 (5.69)
  End of intervention | 26.42 (6.18) | 27.09 (6.09)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in positive mental health across the intervention period; Test type: Superiority; p = .916, Generalized estimating equation; Slope = 0.07, 95% CI 2-sided [-1.17 to 1.30]

19. Secondary Outcome: Changes in Scores on Associated Phenotypes - Stress
Description: Perceived stress, as measured using the Perceived Stress Scale. The theoretical range is 5-50, and a higher score indicates higher levels of perceived stress.
Time Frame: 3 weeks, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Online CBT for Insomnia | Puzzles
Number analyzed (Participants) | 99 | 100
score on a scale
  Mid intervention | 17.92 (8.24) | 19.14 (7.56)
  End of intervention | 16.96 (6.57) | 17.71 (8.06)
Statistical Analysis 1: Comparison: Online CBT for Insomnia vs Puzzles; This analysis looked at the effect of group on changes in perceived stress across the intervention period; Test type: Superiority; p = .027, Generalized estimating equation; Slope = -2.03, 95% CI 2-sided [-3.83 to -0.23]

20. Other Pre Specified Outcome: Online CBT for Insomnia in Sleep Paralysis
Description: Sleep paralysis is a relatively common but understudied phenomenon that has the potential to cause large amounts of fear and/or distress in individuals who experience it. As an exploratory analysis, it shall be investigated whether individuals assigned to the CBT intervention who also experience sleep paralysis show any reductions in the frequency of episodes, and associate levels of fear/distress throughout the programme.
  As this isn't a main aim of the study, this aim is dependent upon a sufficient number of participants who experience sleep paralysis being present in the sample. It is unlikely that there will be sufficient power to thoroughly assess this, but it is hoped this will provide helpful information to future studies.
Time Frame: Change from baseline to 6 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Phenotypic Associations With Exploding Head Syndrome
Description: Exploding head syndrome is an unusual and understudied phenomenon associated with sleep. Measures included in this study shall be used in an exploratory fashion to perform a cross-sectional analysis looking at associations between exploding head syndrome and factors such as sleep problems, depression, anxiety, and well-being.
  Exploding head syndrome was measured using a 1-5 scale, where 1 = never experienced and 5 = several times a week. Sleep paralysis was measured using a 1-7 scale ranging from 1 = never observed to 7 = several times a week.
Time Frame: Baseline
Population: This aim was only focused on the baseline data. Therefore, all participants are included in this analysis independent of which group they were assigned to. As such, results of all participants combined are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: For these analyses, the effect of interest is associations between exploding head syndrome (measured at baseline), and measures of insomnia (Sleep Condition Indicator), anxiety (State/Trait Anxiety Index), depression (Mood and Feelings Questionnaire), stress (Perceived Stress Scale), and sleep paralysis (single item). As such, there is a single obtained value (the regression coefficient + 95% confidence interval).
Arm/Group | All Participants
Number analyzed (Participants) | 199
score on a scale
  Exploding head syndrome | 1.64 (0.98)
  Sleep paralysis | 1.98 (1.35)
Statistical Analysis 1: Comparison: All Participants; Assocation between baseline anxiety symptoms and exploding head syndrome; Test type: Superiority; p = .296, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.77 to 2.40]
Statistical Analysis 2: Comparison: All Participants; Assocation between baseline insomnia symptoms and exploding head syndrome; Test type: Superiority; p = .065, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.47 to 1.02]
Statistical Analysis 3: Comparison: All Participants; Assocation between baseline depression symptoms and exploding head syndrome; Test type: Superiority; p = .145, Regression, Logistic; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.39 to 1.15]
Statistical Analysis 4: Comparison: All Participants; Assocation between baseline life stress and exploding head syndrome; Test type: Superiority; p = .398, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.73 to 2.19]
Statistical Analysis 5: Comparison: All Participants; Assocation between sleep paralysis and exploding head syndrome; Test type: Superiority; p = .001, Regression, Logistic; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.24 to 2.38]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the period of baseline assessments being completed though to the 6-month follow up assessment. This corresponds to a total of 225 days.
Arm/Group | Online CBT for Insomnia | Puzzles
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/100
Other Adverse Events (participants affected / at risk) | 0/99 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT03062891/Prot_SAP_000.pdf